CLINICAL TRIAL: NCT04633291
Title: Clinical Study in Healthy Volunteers Evaluating the Performance and Handling of a Urinary Intermittent Catheter With a Newly Developed Swelling Media.
Brief Title: Investigation of New Intermittent Catheter Swelling Media in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CP279
Record Dates: First submitted 2020-11-05; First posted 2020-11-18 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2022-08

CONDITIONS: Catheter Site Pain; Catheter Site Discomfort

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel swelling media (Experimental): Participants underwent catheterization with the SpeediCath standard male catheter containing the novel swelling media. The catheterization was performed by a trained nurse.
  Interventions: Device: Novel swelling media
- Comparator swelling media (Active Comparator): Participants underwent catheterization with CE-marked SpeediCath® standard male containing the original swelling media. The catheterization was performed by a trained nurse.
  Interventions: Device: Comparator swelling media

INTERVENTIONS:
Device: Novel swelling media — Intermittent catheterization through the urethra draining the bladder, performed by a trained nurse.
  Arms: Novel swelling media
Device: Comparator swelling media — Intermittent catheterization through the urethra draining the bladder, performed by a trained nurse.
  Arms: Comparator swelling media

SUMMARY:
Investigation of novel swelling media for CE marked intermittent urinary catheters. The study was a randomized, single blinded, cross-over investigation comparing a novel swelling media with a comparator swelling media in 22 adult, healthy, male volunteers.

DETAILED DESCRIPTION:
The CP279 study investigated a novel swelling media for male intermittent urinary catheters. The study was conducted in Denmark and was a single-site, randomized, single blinded, cross-over investigation, testing inferiority of a novel catheter swelling media against a comparator swelling media in 22 adult, healthy, male volunteers.

Each participant was randomized to one of two treatment arms, using a randomization sequence of two (i.e., with two different random options for the order in which the participants tested the two swelling media). The study thus contained two test visits, for which the 22 participants tested the two different swelling media, respectively. There was 4-14 days between the test visits and all catheterizations were performed by trained nurses. Due to a visual difference between the products, it was only possible to blind the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent given
* Minimum 18 years of age and with full legal capacity
* Male gender
* Willing to refrain from using analgesics up to 24 hours prior to catheterization visits
* Negative urine multistix analysis for erythrocytes (microscopic hematuria)
* Negative urine multistix analysis for leukocytes and nitrite, or if positive, subsequent negative for bacterial growth in urine culture

Exclusion Criteria:

* Abnormalities, diseases or surgical procedures performed in the lower urinary tract
* Symptoms of urinary tract infections (at least one of the following: frequent urination, stinging or pain at urination)
* Participating in other clinical investigations related to urinary tracts system during this investigation (inclusion to termination) or previously participation in this investigation
* Known hypersensitivity toward any of the investigational device

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Bagi, MD, Principal Investigator — Urologisk klinik Afsnit 2112, Rigshospitalet, Denmark
Locations (1):
- Urologisk klinik Afsnit 2112, Rigshospitalet, Denmark, Copenhagen, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During November 2019, 22 users were recruited for the study from one site (Denmark) and encompassed the safety population.
Pre-assignment Details: The 22 recruited participant were randomized into the two intervention arms, i.e., using a randomization sequence of two. No participants were excluded and none were discontinued.
  Thus, 22 participants constituted the safety and the intention to treat (ITT) population.
Groups:
- Original Swelling Media, Then Novel Swelling Media: On two separate and randomly assigned visits, the participants underwent two interventions:
  First intervention: Day of catheterization with original swelling media (Comparator).
  Washout: 4-14 days. Second intervention: Day of catheterization with novel swelling media (Test device).
- Novel Swelling Media, Then Original Swelling Media: On two separate and randomly assigned visits, the participants underwent two interventions:
  First intervention: Day of catheterization with novel swelling media (Test device).
  Washout: 4-14 days. Second intervention: Day of catheterization with original swelling media (Comparator).
Period: Overall Study
Arm/Group | Original Swelling Media, Then Novel Swelling Media | Novel Swelling Media, Then Original Swelling Media
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total ITT Population: Each treatment arm consisted of two test visits with 4-14 washout days between each crossover. On each visit, the participants underwent intermittent catheterization through the urethra, draining the bladder, and tested a different intermittent catheter: The comparator catheter (SpeediCath® Standard male with original swelling media) or the test catheter (SpeediCath® Standard male with novel swelling media). All catheterizations were performed by a trained nurse.
Arm/Group | Total ITT Population
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 22
Number of participants with presence of hematuria (microscopic) [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Discomfort During Nurse Catheterization
Description: Discomfort measured for the entire catheterization procedure (performed by nurse), using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: The intention to treat population (full analysis set) constituted all randomized subjects with a valid informed consent who was exposed to at least one product, and with valid information on at least one product with respect to the endpoint.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Novel Swelling Media | Comparator Swelling Media
Number analyzed (Participants) | 22 | 22
cm | 1.75 (1.57) | 1.79 (1.86)
Statistical Analysis 1: Comparison: Novel Swelling Media vs Comparator Swelling Media; At a 85% power level, the sample size needed to demonstrate non-inferiority of the novel coating to the original the coating was 18 subjects (participants). This was based on a standard deviation of 1.6 cm, a within subject correlation of 0.5 cm, and an assumption of same VAS distribution for the investigational device as for the comparator. With an expected drop-out rate of 20%, 22 subjects were included; Test type: Non-Inferiority — Based on previous studies, the weighted average VAS discomfort level in healthy subjects using SpeediCath®Standard Male was estimated at 2.3 cm, with 50% increase in VAS was considered clinically relevant. The mean difference non-inferiority margin between catheter coatings was therefore set to 1.2 cm, and non-inferiority was demonstrated if the mean difference was not above 1.2 cm; p = 0.88, Mixed Models Analysis — The threshold for statistical significance was set at 0.05; Random effect: 'Subject'. Fixed effect: 'Visit' (Visit 1 and 2) and 'Treatment' (original coating and novel coating). Age was included as covariate; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.50 to 0.58]

2. Secondary Outcome: Insertion Discomfort During Nurse Catheterization
Description: as for outcome 1
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Novel Swelling Media | Comparator Swelling Media
Number analyzed (Participants) | 22 | 22
cm | 2.17 (1.91) | 2.03 (1.90)
Statistical Analysis 1: Comparison: Novel Swelling Media vs Comparator Swelling Media; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.62, Mixed Models Analysis — The threshold for statistical significance was set at 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.72 to 0.44]

3. Secondary Outcome: Withdrawal Discomfort During Nurse Catheterization
Description: as for outcome 1
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Novel Swelling Media | Comparator Swelling Media
Number analyzed (Participants) | 22 | 22
cm | 1.16 (1.09) | 1.27 (1.37)
Statistical Analysis 1: Comparison: Novel Swelling Media vs Comparator Swelling Media; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.63, Mixed Models Analysis — The threshold for statistical significance was set at 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.36 to 0.57]

4. Secondary Outcome: Urination Discomfort After Catheterization
Description: as for outcome 1
Time Frame: Immediately after first normal void, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Novel Swelling Media | Comparator Swelling Media
Number analyzed (Participants) | 22 | 22
cm | 0.52 (0.71) | 0.37 (0.59)
Statistical Analysis 1: Comparison: Novel Swelling Media vs Comparator Swelling Media; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.19, Mixed Models Analysis — The threshold for statistical significance was set at 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.38 to 0.08]

5. Secondary Outcome: Catheter Handling During Insertion
Description: Nurse evaluation of how he/she experienced catheter insertion on a 5-point likert scale including the options: Very difficult, difficult, neither difficult nor easy, easy or very easy.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Novel Swelling Media | Comparator Swelling Media
Number analyzed (Participants) | 22 | 22
Participants
  Very easy | 8 | 6
  Easy | 7 | 8
  Neither difficult nor easy | 4 | 3
  Difficult | 1 | 4
  Very difficult | 2 | 1
Statistical Analysis 1: Comparison: Novel Swelling Media vs Comparator Swelling Media; Null hypothesis: No difference between the devices; Test type: Superiority; p = 0.381, Proportional odds model — The threshold for statistical significance was set at 0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.47 to 6.60] — OR=1 corresponds to exact equality. OR >1 means that the investigational device is evaluated easier than the comparator. OR <1 means that the comparator device is evaluated easier than the investigational device

6. Secondary Outcome: Catheter Handling During Withdrawal
Description: Nurse evaluation of how he/she experienced catheter withdrawal on a 5-point likert scale including the options: Very difficult, difficult, neither difficult nor easy, easy or very easy.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Novel Swelling Media | Comparator Swelling Media
Number analyzed (Participants) | 22 | 22
Participants
  Very easy | 17 | 13
  Easy | 4 | 8
  Neither difficult nor easy | 0 | 0
  Difficult | 0 | 0
  Very difficult | 1 | 1
Statistical Analysis 1: Comparison: Novel Swelling Media vs Comparator Swelling Media; Null hypothesis: No difference between the devices; Test type: Superiority; p = 0.541, Proportional odds model — The threshold for statistical significance was set at 0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.80, 95% CI 2-sided [-18.40 to 34.00] — OR=1 corresponds to exact equality. OR >1 means that the investigational device is evaluated easier than the comparator. OR <1 means that the comparator device is evaluated easier than the investigational device. Of note: Log transformed estimates

7. Secondary Outcome: Touch of Catheter Coating
Description: Nurse evaluation of whether or not it was needed to touch the catheter coating during handling and/or catheterization (yes/no).
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Novel Swelling Media | Comparator Swelling Media
Number analyzed (Participants) | 22 | 22
Participants
  Yes | 4 | 3
  No | 18 | 19
Statistical Analysis 1: Comparison: Novel Swelling Media vs Comparator Swelling Media; Null hypothesis: No difference between the devices; Test type: Superiority; p = 0.269, Regression, Logistic — The threshold for statistical significance was set at 0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.17, 95% CI 2-sided [0.19 to 265.95] — OR=1 corresponds to exact equality. OR >1 means that the investigational device is in favor compared to the comparator. OR <1 means that the comparator device is in favor compared to the investigational device

8. Secondary Outcome: Visual Blood During Catheterization
Description: Nurse evaluation of if he/she experienced visual blood on either the catheter or in the urine during catheterization (yes/no).
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Novel Swelling Media | Comparator Swelling Media
Number analyzed (Participants) | 22 | 22
Participants
  Yes | 1 | 1
  No | 21 | 21
Statistical Analysis 1: Comparison: Novel Swelling Media vs Comparator Swelling Media; Null hypothesis: No difference between the devices; Test type: Superiority; p = 1.0, Regression, Logistic — The threshold for statistical significance was set at 0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.02 to 64.83] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Microscopic Blood in Catheter-collected Urine
Description: Dipstick analysis of hematuria (erythrocytes) after catheterization using a semi-quantitative color scale with five categories ranging from negative to 3+:
  Negative (-). 10 erythrocytes/μL (+/-). 25 erythrocytes/μL (1+). 80 erythrocytes/μL (2+). 200 erythrocytes/μL (3+).
  At least one fully positive response (i.e., either 1+, 2+ or 3+), the endpoint was considered positive and the outcome was analyzed as a binary response (positive/negative).
Time Frame: Immediately after the procedure/catheterization, up to 30 min.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Novel Swelling Media | Comparator Swelling Media
Number analyzed (Participants) | 22 | 22
Participants
  Hematuria positive | 6 | 6
  Hematuria negative | 16 | 16
Statistical Analysis 1: Comparison: Novel Swelling Media vs Comparator Swelling Media; Null hypothesis: No difference between the devices; Test type: Superiority; p = 1.0, Regression, Logistic — The threshold for statistical significance was set at 0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.08 to 12.87] — [estimate comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: Each participant was enrolled for 5-15 days for the entire investigation, thus a maximum of 15 days.
Description: The relationship to the investigational or comparator products was collected. The safety population constituted the subjects who had given informed consent and were thus 22 participants.
  An adverse event was reported as either: "Not related", "Unlikely related", "Possibly related", "Probably related", or "Definitely related", to the intervention.
Arm/Group | Novel Swelling Media | Comparator Swelling Media
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT04633291/Prot_SAP_000.pdf